CLINICAL TRIAL: NCT01395602
Title: Randomized Controlled Pilot Study of the Effect of Cabergoline on Body Weight and Glucose Tolerance in Healthy Obese Adults
Brief Title: Effect of Cabergoline on Weight and Glucose Tolerance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Judith Korner, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IRB #13952
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Body Weight; Impaired Glucose Tolerance in Obese
MeSH Terms: conditions — Body Weight | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo pill
  Interventions: Other: placebo
- cabergoline (Active Comparator): cabergoline pill
  Interventions: Drug: Cabergoline

INTERVENTIONS:
Drug: Cabergoline — cabergoline 0.5 mg twice weekly
  Arms: cabergoline
Other: placebo — 1 pill twice weekly
  Arms: placebo

SUMMARY:
The aim of this study is to determine the efficacy of cabergoline, a long-acting dopamine receptor agonist, on body weight and blood glucose in healthy obese adults.

This is a randomized double-blind placebo controlled study. Twenty subjects each will be randomly assigned either placebo or cabergoline for 16 weeks.

The effect of treatment on body weight and blood glucose and insulin levels will be compared in the treatment versus the placebo arm.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 55 years
* BMI 30 -40

Exclusion Criteria:

* diabetes,
* clinically significant medical condition,
* use of medications that effect blood glucose or body weight

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2002-04; Primary Completion 2003-09 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
body weight | 16 weeks

SECONDARY OUTCOMES:
glucose | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judith Korner, MD, PHD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States